CLINICAL TRIAL: NCT00751114
Title: Superiority Study of Insulin Glargine Over Sitagliptin in Insulin-naïve Patients With Type 2 Diabetes Treated With Metformin and Not Adequately Controlled
Brief Title: Evaluation of Insulin Glargine Versus Sitagliptin in Insulin-naive Patients
Acronym: EASIE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_C_02761; 2008-000516-32 (EudraCT Number)
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Results first posted 2012-08-15 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Sitagliptin Phosphate; Metformin

ARMS (2):
- Insulin Glargine (Experimental): Administered once a day in the evening at dinner or at bedtime with a starting dose 0.2 U/kg. Then, the doses were to be individually adjusted, following a titration algorithm, to reach the FPG target: 70mg/dL<FPG≤100mg/dL (3.9mmol/L<FPG≤5.5mmol/L).
  Interventions: Drug: Insulin Glargine; Drug: Metformin
- Sitagliptin (Active Comparator): Dose of 100 mg once a day administered with or without food.
  Interventions: Drug: Sitagliptin; Drug: Metformin

INTERVENTIONS:
Drug: Insulin Glargine — Subcutaneous injection. 100 Units/mL solution for injection in a pre-filled SoloStar® pen (3 mL).
  Other Names: Lantus®
  Arms: Insulin Glargine
Drug: Sitagliptin — Oral administration. 100 mg film-coated tablets.
  Other Names: Januvia®
  Arms: Sitagliptin
Drug: Metformin — Patients continued with metformin as usual oral anti-diabetic treatment.

SUMMARY:
The primary objective was to demonstrate the superiority of insulin glargine over sitagliptin in reducing Glycosylated Hemoglobin A1c (HbA1c) from baseline to the end of the treatment period.

Secondary objective was to assess the effect of insulin glargine in comparison with sitagliptin on:

* HbA1c level
* Fasting Plasma Glucose (FPG)
* 7-point plasma glucose (PG) profiles
* Percentage of patients with HbA1c <7% and <6.5%

Safety objectives consisted of:

* Hypoglycemia occurrence
* Body weight
* Overall safety

ELIGIBILITY:
Inclusion Criteria:

* With type 2 diabetes diagnosed for at least 6 months,
* Not previously treated with insulin,
* On metformin for at least 3 months and a stable minimal dose of 1 g/day for at least 2 months
* HbA1c ≥ 7 and < 11 %,
* Body Mass Index (BMI) between 25 and 45 kg/m² inclusively,
* Ability and willingness to perform plasma glucose (PG) monitoring using the Sponsor-provided PG meter and to complete the patient diary,
* Signed informed consent obtained prior any study procedures,
* Willingness and ability to comply with the study protocol.

Exclusion Criteria:

* Treatment with oral antidiabetic drugs other than metformin within the last 3 months,
* Previous treatment with the combination of metformin + sulfonylurea for more than 1 year,
* Previous treatment with Glucagon Like Peptide-1 (GLP-1) agonists or DiPeptidyl Peptidase (DPP) IV inhibitors,
* FPG (assessed by central laboratory measurement) ≥ 280 mg/dL (15.4 mmol/L),
* Diabetes other than type 2 diabetes (e.g. secondary to pancreatic disorders, drug or chemical agents intake...),
* Pregnant or lactating women (women of childbearing potential must have a negative pregnancy test at study entry and a medically approved contraception method),
* In-patient care,
* Active proliferative retinopathy, as defined by a photocoagulation or vitrectomy occurrence in the 6 months prior to visit 1, or any other unstable (rapidly progressing) retinopathy that may require photocoagulation or surgical treatment during the study (an optic fundus examination should have been performed within the 2 years prior to study entry),
* Impaired renal function: serum creatinine ≥ 1.5 mg/dL (≥ 133µmol/L) or ≥ 1.4 mg/dL (≥ 124 µmol/L) in men and women, respectively,
* History of sensitivity to the study drugs or to drugs with a similar chemical structure,
* Impaired hepatic function: alanine aminotransferase (ALT), aspartate aminotransferase (AST) > 3 x upper limit of normal range,
* Treatment with systemic corticosteroids within the 3 months prior to study entry or likelihood of requiring treatment during the study that are not permitted during the study (exception: in case of chronic adrenal insufficiency, systemic glucosteroids are accepted only if the disease is stable and the treatment dose stable for at least 3 months before study entry),
* Alcohol or drug abuse within the last year,
* Night shift worker,
* Presence of any condition (medical, psychological, social or geographical), current or anticipated that the investigator feels would compromise the patient's safety or limit the patient successful participation in the study,
* Treatment with weight loss medications (e.g. sibutramine, orlistat, rimonabant) within the last 3 months,
* Participation in another clinical trial within the month prior to visit 1,
* History of pancreatitis.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2008-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (17):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Cairo, Egypt
- Sanofi-Aventis Administrative Office, Kallithea, Greece
- Sanofi-Aventis Administrative Office, Hong Kong, Hong Kong
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Beirut, Lebanon
- Sanofi-Aventis Administrative Office, Col. Coyoacan, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Result] Aschner P, Chan J, Owens DR, Picard S, Wang E, Dain MP, Pilorget V, Echtay A, Fonseca V; EASIE investigators. Insulin glargine versus sitagliptin in insulin-naive patients with type 2 diabetes mellitus uncontrolled on metformin (EASIE): a multicentre, randomised open-label trial. Lancet. 2012 Jun 16;379(9833):2262-9. doi: 10.1016/S0140-6736(12)60439-5. Epub 2012 Jun 9. PMID 22683131
- [Derived] Chan JC, Aschner P, Owens DR, Picard S, Vincent M, Dain MP, Pilorget V, Loizeau V, Echtay A, Fonseca V. Triple combination of insulin glargine, sitagliptin and metformin in type 2 diabetes: the EASIE post-hoc analysis and extension trial. J Diabetes Complications. 2015 Jan-Feb;29(1):134-41. doi: 10.1016/j.jdiacomp.2014.08.007. Epub 2014 Aug 27. PMID 25283485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: EASIE was a multicenter, international, randomized, open-label trial conducted from November 12, 2008 to July 28, 2011.
Pre-assignment Details: A total of 732 patients were screened in 96 centers in 17 countries. The study included an initial 2-week screening period. A total of 217 patients were screen failures. The main reason for screen failure was Glycosylated Hemoglobin A1c (HbA1c) inclusion criterion not met (146 patients).
Groups:
- Insulin Glargine: Administered once a day in the evening at dinner or at bedtime with a starting dose 0.2 U/kg. Then, the doses were to be individually adjusted, following a titration algorithm, to reach the Fasting Plasma Glucose (FPG) target: 70mg/dL<FPG≤100mg/dL (3.9mmol/L<FPG≤5.5mmol/L)
Period: Overall Study
Arm/Group | Insulin Glargine | Sitagliptin
Started | 250 (randomized) | 265
TREATED = Safety Population | 237 (safety population: randomized patients who received at least one dose of investigational product) | 264
mITT Population | 227 (modified Intent-To-Treat population: treated patients with at least 1 on-treatment efficacy measure) | 253
Completed | 212 | 233
Not Completed | 38 | 32
Not completed — Adverse Event | 2 | 4
Not completed — Protocol Violation | 8 | 9
Not completed — Withdrawal by Subject | 9 | 4
Not completed — Lost to Follow-up | 4 | 7
Not completed — Lack of Efficacy | 0 | 7
Not completed — Not Treated | 13 | 1
Not completed — Out of country for 2 months | 1 | 0
Not completed — Move to another city | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Glargine | Sitagliptin | Total
Number analyzed (Participants) | 227 | 253 | 480
Age Continuous [Mean (Standard Deviation); unit: years] — mITT population
  years | 53.9 (8.9) | 53.3 (8.7) | 53.6 (8.8)
Sex/Gender, Customized [Number; unit: participants] — mITT population
  participants
    Male | 114 | 132 | 246
    Female | 113 | 121 | 234
Body Weight [Mean (Standard Deviation); unit: kg] — mITT population
  kg | 83.4 (18.2) | 84.2 (18.3) | 83.8 (18.2)
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] — mITT population
  kg/m² | 31.05 (4.93) | 31.13 (4.95) | 31.09 (4.93)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — mITT population
  mmHg | 129.8 (13.3) | 131.7 (15.1) | 130.8 (14.3)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — mITT population
  mmHg | 79.5 (8.7) | 80.0 (8.3) | 79.7 (8.5)
Heart Rate [Mean (Standard Deviation); unit: beats/min] — mITT population
  beats/min | 75.6 (8.7) | 76.3 (9.3) | 76.0 (9.0)
Duration of diabetes [Median (Inter-Quartile Range); unit: years] — mITT population
  years | 3.9 [1.9 to 8.2] | 4.8 [1.9 to 8.2] | 4.5 [1.9 to 8.2]
At least one diabetic late complication [Number; unit: participants] — mITT population
  Diabetic late complications: myocardial infarction, angina pectoris, coronary artery disease, heart failure, stroke, transient ischemic attack, peripheral vascular disease, diabetic neuropathy, diabetic nephropathy, diabetic retinopathy
  participants
    Yes | 65 | 67 | 132
    No | 162 | 186 | 348
Glycosylated Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percent] — mITT population
  percent | 8.5 (1.0) | 8.5 (1.1) | 8.5 (1.1)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] — mITT population but due to missing values, N=225 for Insulin Glargine and N=248 for Sitagliptin
  mg/dL | 163.6 (42.0) | 171.1 (41.5) | 167.5 (41.9)
Self-monitored Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] — mITT population but due to missing values, N=216 for Insulin Glargine and N=244 for Sitagliptin
  mg/dL | 163.9 (37.6) | 166.7 (38.2) | 165.4 (37.9)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] — mITT population but due to missing values, N=225 for Insulin Glargine and N=248 for Sitagliptin
  mg/dL | 185.9 (41.4) | 187.1 (39.0) | 186.5 (40.1)
High-Density Lipoprotein (HDL) Cholesterol [Mean (Standard Deviation); unit: mg/dL] — mITT population but due to missing values, N=225 for Insulin Glargine and N=248 for Sitagliptin
  mg/dL | 46.2 (14.6) | 45.0 (11.2) | 45.6 (12.9)
Low-Density Lipoprotein (LDL) Cholesterol [Mean (Standard Deviation); unit: mg/dL] — mITT population but due to missing values, N=225 for Insulin Glargine and N=248 for Sitagliptin
  mg/dL | 112.7 (36.2) | 114.2 (33.2) | 113.5 (34.6)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] — mITT population but due to missing values, N=225 for Insulin Glargine and N=248 for Sitagliptin
  mg/dL | 190.9 (142.0) | 185.7 (114.6) | 188.2 (128.3)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c: Change From Baseline to Study Endpoint
Description: Change in HbA1c from baseline to study endpoint defined as the last available HbA1c value measured during the 24-week treatment period.
Time Frame: baseline (week 0), study endpoint: visit 14 (week 24) or visit 11 (week 12) if value not available at visit 14
Population: The population analyzed for this outcome measure consisted of the subset of mITT patients who had both baseline and endpoint measurements.
  The Last Observation Carried Forward method was used for imputing missing data for the end of treatment value.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Insulin Glargine | Sitagliptin
Number analyzed (Participants) | 224 | 248
percent | -1.72 (0.06) | -1.13 (0.06)
Statistical Analysis 1: Comparison: Insulin Glargine vs Sitagliptin; H0: no difference between insulin glargine mean HbA1c change and sitagliptin mean HbA1c change H1: difference between insulin glargine mean HbA1c change and sitagliptin mean HbA1c change Assuming: * Estimated standard deviation of the change in HbA1c of 1.3% * Expected mean difference to be detected of 0.4% * Alpha risk of 5% (two-sided) * Power of 90% * Equal sample size in each treatment group (1:1 randomization) A total number of 446 evaluable patients (223 in each group) was required; Test type: Superiority or Other; p < 0.0001, ANCOVA — An analysis of covariance (ANCOVA) was performed, with the HbA1c change from baseline to last on-treatment measurement as dependent variable, treatment as fixed effect and the corresponding baseline HbA1c value as covariate; adjusted mean difference = -0.59, 95% CI 2-sided [-0.77 to -0.42], Standard Error of Mean 0.09 — Difference (Insulin glargine - Sitagliptin)

2. Secondary Outcome: HbA1c Response Rate: Percentage of Patients Who Reach the Target of HbA1c < 7% at Study Endpoint
Time Frame: study endpoint: visit 14 (week 24) or visit 11 (week 12) if value not available at visit 14
Population: The population analyzed for this outcome measure consisted of the subset of mITT patients who had endpoint measurements.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Sitagliptin
Number analyzed (Participants) | 224 | 248
percentage of participants | 67.9 | 41.9

3. Secondary Outcome: HbA1c Response Rate: Percentage of Patients Who Reach the Target of HbA1c < 6.5% at Study Endpoint
Time Frame: study endpoint: visit 14 (week 24) or visit 11 (week 12) if value not available at visit 14
Population: The population analyzed for this outcome measure consisted of the subset of mITT patients who had endpoint measurements.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Sitagliptin
Number analyzed (Participants) | 224 | 248
percentage of participants | 40.2 | 16.9

4. Secondary Outcome: Self-monitored Fasting Plasma Glucose (SMFPG) Mean : Change From Baseline to Study Endpoint
Description: SMFPG mean = mean of the fasting plasma glucose values recorded on the 6 consecutive days before the visit (at least 3 values needed).
  Study endpoint was defined as the last available SMFPG mean value collected on-treatment.
  Change= study endpoint - baseline
Time Frame: baseline (week 0), study endpoint: visit 14 (week 24) or visit 12 (week 16) or visit 11 (week 12) or visit 8 (week 6) depending on last available value
Population: The population analyzed for this outcome measure consisted of the subset of mITT patients who had both baseline and endpoint measurements.
  Adjusted means were estimated from ANCOVA model using baseline value as covariate.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Glargine | Sitagliptin
Number analyzed (Participants) | 214 | 244
mg/dL | -60.52 (1.85) | -19.35 (1.73)

5. Secondary Outcome: 7-point Plasma Glucose Profile: Change From Baseline to Study Endpoint
Description: 7-point plasma glucose recorded before and after breakfast, before and after lunch, before and after dinner and at bedtime.
  Change = study endpoint - baseline.
Time Frame: baseline (week 0), study endpoint: visit 14 (week 24) or visit 11 (week 12) if value not available at visit 14
Population: The population analyzed for this outcome measure consisted of the subset of mITT patients who had valid 7-point plasma glucose profiles (4 points needed for a valid profile) both at baseline and endpoint.
  Depending on the time point, few values were missing.
  Adjusted means were estimated from ANCOVA model using baseline value as covariate.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Glargine | Sitagliptin
Number analyzed (Participants) | 203 | 227
mg/dL
  Before breakfast (N ig = 203 & N s = 226) | -59.90 (2.02) | -20.39 (1.91)
  After breakfast (N ig = 202 & N s = 220) | -66.25 (3.03) | -36.41 (2.90)
  Before lunch (N ig = 201 & N s = 223) | -48.00 (2.33) | -19.82 (2.21)
  After lunch (N ig = 202 & N s = 226) | -45.54 (2.82) | -26.10 (2.66)
  Before dinner (N ig = 199 & N s = 223) | -40.68 (2.61) | -25.07 (2.47)
  After dinner (N ig = 196 & N s = 220) | -45.88 (2.69) | -33.78 (2.54)
  At bedtime (N ig = 177 & N s = 210) | -45.58 (3.15) | -31.16 (2.89)

6. Secondary Outcome: Insulin Dose in the Insulin Glargine Group
Description: Daily dose at the face-to-face visits.
Time Frame: visit 4 (week 2), visit 8 (week 6), visit 11 (week 12), visit 12 (week 16), visit 14 (week 24), first dose received defined as first available value, study endpoint defined as last available value
Population: The population analyzed for this outcome was the safety population defined as randomized patients who received at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: unit per kg body weight
Arm/Group | Insulin Glargine
Number analyzed (Participants) | 237
unit per kg body weight
  First dose received N=236 | 0.19 (0.03)
  Visit 4 (week 2) N=230 | 0.27 (0.08)
  Visit 8 (week 6) N=222 | 0.38 (0.16)
  Visit 11 (week 12) N=219 | 0.45 (0.20)
  Visit 12 (week 16) N=214 | 0.48 (0.23)
  Visit 14 (week 24) N=220 | 0.50 (0.26)
  Study endpoint N=237 | 0.49 (0.26)

7. Secondary Outcome: Lipid Profile: Change From Baseline to Study Endpoint
Time Frame: baseline (week 0), study endpoint: visit 14 (week 24) or visit 11 (week 12) if value not available at visit 14
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Glargine | Sitagliptin
Number analyzed (Participants) | 222 | 243
mg/dL
  Change in Total Cholesterol | -7.94 (2.06) | -1.54 (1.97)
  Change in LDL Cholesterol | -3.68 (1.71) | -0.19 (1.63)
  Change in HDL Cholesterol | 0.13 (0.54) | 0.57 (0.52)
  Change in Triglycerides | -34.07 (8.14) | 0.31 (7.78)

8. Secondary Outcome: Change in Body Weight From Baseline to Study Endpoint
Time Frame: as for outcome 4
Population: The population analyzed for this outcome measure consisted of the subset of the safety population (treated patients) who had both baseline and endpoint measurements.
  Adjusted means were estimated from ANCOVA model using baseline value as covariate.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Insulin Glargine | Sitagliptin
Number analyzed (Participants) | 227 | 255
kg | 0.44 (0.22) | -1.08 (0.20)

9. Secondary Outcome: Number of Patients With at Least One Episode of Symptomatic Hypoglycemia
Description: Symptomatic hypoglycemia was defined as an event with clinical symptoms that were considered to result from hypoglycemia confirmed or not by a plasma glucose measurement <= 70mg/dL [3.9 mmol/L]
Time Frame: During the treatment phase (24 weeks) plus 7 days after last dose
Population: The population analyzed for this outcome measure was the safety population (treated patients)
Measure: Number; unit: participants
Arm/Group | Insulin Glargine | Sitagliptin
Number analyzed (Participants) | 237 | 264
participants | 108 | 35

10. Secondary Outcome: Number of Patients With at Least One Episode of Severe Symptomatic Hypoglycemia
Description: Severe symptomatic hypoglycemia was defined as an event with clinical symptoms which required assistance of another person and with either a Plasma Glucose level < 36 mg/dL (2 mmol/L) or with a prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration
Time Frame: During the treatment phase (24 weeks) plus 7 days after last dose
Population: The population analyzed for this outcome measure was the safety population (treated patients)
Measure: Number; unit: participants
Arm/Group | Insulin Glargine | Sitagliptin
Number analyzed (Participants) | 237 | 264
participants | 3 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were assessed throughout the study (24 weeks). Mean duration of exposure to insulin glargine was 157.7 ± 40.9 days (ranging from 1 to 211 days) and 160.8 ± 33.7 days to sitagliptin (ranging from 14 to 262 days).
Arm/Group | Insulin Glargine | Sitagliptin
Serious Adverse Events (participants affected / at risk) | 15/237 | 8/264
Other Adverse Events (participants affected / at risk) | 27/237 | 41/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin Glargine (N=237) | Sitagliptin (N=264)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 2 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin Glargine (N=237) | Sitagliptin (N=264)
Influenza (Infections and infestations) | 8 | 15
Nasopharyngitis (Infections and infestations) | 8 | 15
Headache (Nervous system disorders) | 15 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 45 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.